CLINICAL TRIAL: NCT00062816
Title: Addition of ISIS 14803 to Therapy With Peginterferon and Ribavirin for Chronic Hepatitis C (HCV) Patients Not Responding Adequately to the Two Drugs
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ISIS 14803-CS3
Record Dates: First submitted 2003-06-16; First posted 2003-06-18 (Estimated); Last update posted 2022-12-05 (Actual); Status verified 2007-10

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis; Chronic
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis; Bronchiolitis Obliterans Syndrome | interventions — Ribavirin

INTERVENTIONS:
Drug: ISIS 14803, peginterferon alfa, ribavirin

SUMMARY:
The purposes of this Phase 1/2 study are to examine the safety, tolerability, and antiviral activity of ISIS 14803, when given in combination with peginterferon alfa and ribavirin, to patients who either failed to have at least a 100-fold HCV reduction at Week 12 of standard therapy or still have detectable HCV at Week 24.

DETAILED DESCRIPTION:
Previously untreated chronic hepatitis C patients undergoing therapy with peginterferon alfa and ribavirin have a very poor probability of achieving a sustained virologic response if they either do not have a 100-fold or greater reduction in their plasma HCV RNA levels at the 12th week of treatment or have detectable plasma HCV RNA at the 24th week of treatment. ISIS 14803 is an experimental antiviral medication for the treatment of chronic hepatitis C that has been given to chronic hepatitis C patients in two previous single-agent clinical trials (approximately 70 patients).

In this clinical research study, 12 weeks of ISIS 14803 treatment will be added to the peginterferon alfa and ribavirin treatment regimen of previously untreated chronic hepatitis C patients who have a very poor probability of achieving a sustained virologic response based upon either of the above two criteria. Enrolled patients must continue to be treated with peginterferon alfa and ribavirin and must begin ISIS 14803 treatment within four weeks of their HCV RNA result report date. ISIS 14803 will be given as a two-hour intravenous infusion, two times each week, for 12 weeks. Depending on their HCV response to the three-drug combination, patients may continue treatment with peginterferon alfa and ribavirin after the end of ISIS 14803 treatment. Patients will be monitored for at least eight weeks (for safety) after the end of ISIS 14803 treatment and possibly for longer (for sustained virologic response). Two dose levels of ISIS 14803 will be studied in this trial, 3 and 6 mg/kg ideal body weight.

ELIGIBILITY:
Inclusion Criteria (partial list):

* Age 18 to 65 years.
* Infection with HCV.
* Prior liver biopsy indicating chronic hepatitis.
* Received at least 12 weeks of continuous peginterferon alfa and ribavirin therapy.
* HCV infection was untreated prior to current peginterferon alfa and ribavirin regimen.
* Either less than 100-fold reduction in plasma or serum HCV RNA despite receiving 12 weeks of peginterferon alfa and ribavirin therapy or detectable HCV RNA at week 24 of therapy.
* Prothrombin time and aPTT within normal reference range.
* Serum bilirubin concentration within normal reference range.
* Give written informed consent to participate in the study.

Exclusion criteria (partial list):

* Pregnant women or nursing mothers or women of childbearing potential without adequate contraception.
* Systemic corticosteroid therapy within 3 months of screening.
* Serum ALT greater than 5 x upper limit of normal range.
* HIV or HBV infection.
* Decompensated liver disease.
* Evidence of cirrhosis.
* Severe depression with suicidal ideation requiring hospitalization within one year of screening.
* Any disease condition associated with active bleeding or requiring anticoagulation with heparin or warfarin.
* Any condition which, in the opinion of the Investigator, would preclude participation in or interfere with compliance.
* Alcohol or drug abuse.
* Is undergoing or has undergone treatment with another investigational drug, biologic agent or device within 30 days of screening
* History of cryoglobulinemia or vasculitis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22
Dates: Start 2003-06; Primary Completion 2004-01 (Actual); Study Completion 2004-01

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - Birmingham Gastroenterology Associates, Birmingham, Alabama
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Community Clinical Trials, Orange, California
  - The Lynn Institute of the Rockies, Colorado Springs, Colorado
  - Western States Clinical Research, Inc., Wheat Ridge, Colorado
  - University of Florida, Jacksonville, Florida
  - Miami Research Associates, Inc., Miami, Florida
  - Idaho Gastroenterology Assoc., Boise, Idaho
  - IMG Healthcare, LLC, New Orleans, Louisiana
  - Beth Israel Deconess Medical Center, Boston, Massachusetts
  - FutureCare Studies, Springfield, Massachusetts
  - William Beaumont Hospital, Royal Oak, Michigan
  - Saint Louis University, St Louis, Missouri
  - Cornell Medical Center, New York, New York
  - Rochester Institute for Digestive Diseases and Sciences, Inc., Rochester, New York
  - Duke Clinical Research Institute, Durham, North Carolina
  - Consultants for Clinical Research, Cincinnati, Ohio
  - Blair Gastroenterology Associates, Altoona, Pennsylvania
  - Gastroenterology Center of the MidSouth, P.C., Germantown, Tennessee
  - Memphis Gastroenterology Group, Memphis, Tennessee
  - Nashville Medical Research Institute, Nashville, Tennessee
  - Baylor College of Medicine-VAMC, Houston, Texas
  - McGuire VAMC, Richmond, Virginia
  - Northwest Gastroenterolgy Assoc., Bellevue, Washington
  - Spokane Digestive Disease Center, Spokane, Washington